CLINICAL TRIAL: NCT04953377
Title: Pelvic Floor Muscle Training Educational Intervention for Patients With Breast Cancer
Brief Title: PFMT Educational Intervention for Patients With Advancer Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Onkologikoa (Other)
Responsible Party: Principal Investigator, Mireia Peláez Puente, PhD, Onkologikoa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onkologikoa
Record Dates: First submitted 2021-06-25; First posted 2021-07-08 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Advanced Breast Cancer
Keywords: pelvic floor muscle training; urinary incontinence; educational intervention
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): PFMT educational intervention including a 120 min workshop and 8 weeks of self training
  Interventions: Behavioral: PFMT educational intervention

INTERVENTIONS:
Behavioral: PFMT educational intervention — an educational intervention to learn about the pelvic floor and how to train it

SUMMARY:
A PFMT educational intervention was designed for women with metastasic breast cancer. It consisted in a 120 min workshop and 8 weeks of non-supervised (but with follow-up) self-training. ICIQ, IQOL and ad hoc questions were performed before the workshop and after the 8 weeks training to see the prevalence of UI, the impact in their quality of life and the empowerment of self-training.

DETAILED DESCRIPTION:
Urinary incontinence (UI) affects women of all ages and has a great impact on the quality of life. Cancer treatments such as chemotherapy or hormone therapy may play an important rol in the development and worsening of pelvic floor disorders. Little evidence on the prevalence and impact of UI in metastassis breast cancer women is known.

A protocol was designed to analyze the effect of a PFMT educational intervention on the UI and the impact on the QoL, as well as in the empowerment feeling of the participants. Feasibility of the protocol will be analized to design an optimal RCT for testing our hypothesis

During the usual visits, oncologist wil recruit women with advanced breast cancer who meet the inclusion criteria for the participation.

ELIGIBILITY:
Inclusion Criteria:

* Advanced breast cancer
* Over 18 years old
* ECOG≤2
* No inestable bone metastasis
* life expentancy>6 months
* Literate in spanish

Exclusion Criteria:

* Physical exercise contraindications
* Intense pain
* Being pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility- Recruitment rates | 8 weeks
  Number of patients enrolled divided by number of patients eligible
Feasibility - Qualitative analyses of recruitment | 8 weeks
  Qualitative information regarding recruitment and reasons for patients not participating will be collected in the researchers log
Feasibility-Quantitative and qualitative retention log | 8 weeks
  Information about number of participants who dropped out, and reason for drop-out
Feasibility- Adherence to the program | 8 weeks
  Adherence will be difined as the percentage of completed weeks of training out of 8 weeks. A week will be considerered valid when the train was performed at least in 2 different days.
Feasibility- Satisfaction with the workshop | baseline
  A satisfaction 9 item questionnaire was design (Scale 1-5) to obtain information about the satisfaction with the (1) duration, (2) the content, (3) explanations, (4) atmosphere (5)number of participants during the workshop and (6) the importance for other patients to access this information, (7) increase in knowledge, (8) knowledge to train alone and (9) overall satisfaction.
Prevalence of urinary incontinence | baseline
  By the ICIQ-UI Short Form, which is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. It has 4 items, and the scoring scale is 0-21.

SECONDARY OUTCOMES:
Changes in urinary incontinence | 8 weeks
  By the ICIQ-UI Short Form, which is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. It has 4 items, and the scoring scale is 0-21.
Impact of urinary incontinence on the quality of life | 8 weeks
  The I-QOL measures the effect of urinary incontinence on quality of life.It is divided into 3 subscales: Avoidance and limiting behavior, Psychosocial impact, and Social embarrassment (SE). Subjects use a 5-point response scale with values ranging from 1 (extremely) to 5 (not at all)
Knowledge and empowerment | 8 weeks
  A 11 item questionnaire was designed to analyse the population's initial knowledge of pelvic floor health and compare it with the knowledge maintained after the intervention. 5-point scale (0-4).

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Pelaez, Principal Investigator — Onkologikoa
Locations (1):
- Onkologikoa, San Sebastián, Spain

IPD SHARING:
Plan to Share IPD: No